CLINICAL TRIAL: NCT04521699
Title: Examination of the Impact of CalmiGo's Stress Management Device on Vascular Health and Cardiovascular Disease Risk , and Markers of Mental Stress in Patients Following a Myocardial Infarction Participating in Clinically Indicated Cardiac Rehabilitation
Brief Title: Examination of the Impact of CalmiGo's Stress Management Device on Vascular Heath and Cardiovascular Disease Risk.
Acronym: CalmiGo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: CalmiGO (Unknown)
Responsible Party: Principal Investigator, Amir Lerman, Dr. Amir Lerman, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-005047
Record Dates: First submitted 2020-08-19; First posted 2020-08-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CalmioGo + Standard of care (Experimental): Use of CalmiGO stress management device once daily + standard of care during the 12 weeks of Cardiac rehabilitation
  Interventions: Device: CalmioGO Stress management device
- Standard of Care (No Intervention): Stand of care alone with 12 weeks of Cardiac rehabilitation

INTERVENTIONS:
Device: CalmioGO Stress management device — CalmiGo device is a device of similar size to an inhaler that uses guided breathing, and grounding techniques to regulate breathing to bring users a sense of calm and relaxation.
  Arms: CalmioGo + Standard of care

SUMMARY:
The primary purpose of this study is to determine if there are significant differences with respect to baseline between those randomized to CGo and standard-of-care versus standard-of-care alone after completing 12-weeks of therapy in terms of peripheral endothelial function measured by EndoPAT.

DETAILED DESCRIPTION:
100 patients who have recently had an acute Myocardial Infarction ( heart attack) and are under going clinically indicated cardiac rehabilitation will undergo baseline testing including EndoPAT testing, mental stress testing, blood tests for cardiovascular disease biomarkers , physical assessments & survey questionnaires. Patients then will be randomized to either CalmioGO stress management device + standard of care treatment or just standard of care treatment. Those randomized to CalmiGO stress management device treatment will be instructed to use the hand device much like an inhaler once a day for 12 weeks. After 12 weeks of rehabilitation both groups will return for reassessment of baseline tests.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ability to use the CamliGo device for 12-weeks
* Willingness to complete study questionnaires, blood tests,& EndoPat testing at the beginning and end of study
* Patients who have had a recent MI who will be undergoing clinically indicated Cardiac Rehabilitation
* Patients who have had a coronary or structural intervention performed in the cardiac catheterization laboratory within the last month, including: coronary stenting; coronary balloon angioplasty; transcatheter aortic valve replacement; mitral valve interventions; patent foramen ovale closures; alcohol septal ablation; paravalvular leak closure.
* Patients being seen in the Chest Pain Clinic for Atypical chest pain

Exclusion Criteria:

* Cognitively impaired patients
* Patient with Bipolar disorder, psychosis or delusional disorder
* History of substance abuse or dependence
* History of suicidality
* Unstable cardiovascular or pulmonary disease
* History of seizures
* Latex allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Peripheral endothelial function | 16 weeks
  Measurements made at baseline will be significantly different between those randomized to CalmioGo + standard of care to those receiving only standard of care treatment

SECONDARY OUTCOMES:
Physical assessments, cardiovascular disease biomarker blood tests as well resilience, joy, gratitude, mindfulness, health behavior , overall quality of life & perceived stress. | 16 weeks
  Measurements made at baseline will be significantly different between those randomized to CalmiGo + standard of care then those to just standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No